CLINICAL TRIAL: NCT06847282
Title: Motor Outcomes to Validate Evaluations in Pediatric FSHD (MOVE Peds)
Acronym: MOVE Peds
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Rochester (Other); Stanford University (Other); Duke University (Other); University of California, Irvine (Other); Kennedy Krieger Institute, Baltimore, MD (Unknown); University of Utah (Other); Seattle Children's Hospital (Other); University of Iowa (Other); Coriell Institute (Unknown); Leiden University Medical Center (Other); Murdoch Childrens Research Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Statland, Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160879; 1U01NS137702-01 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-02-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: FSHD; Pediatric
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be collected at baseline for genetic testing and will be sent to Leiden for assessment. DNA, plasma, and serum biomarker samples that are collected will be sent to Coriell which will be stored in a biorepository for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort One: Cohort One will be individuals who are able to complete the 10 meter walk/run test in less than twelve seconds
- Cohort Two: cohort two will be individuals who complete the 10 meter walk/run test in more than 12 seconds or is no longer able to complete.

SUMMARY:
The primary goal of this study is to validate motor and functional outcomes and refine clinical trial strategies for pediatric-onset FSHD

DETAILED DESCRIPTION:
MOVE Peds is a prospective 2-year study recruiting eighty pediatric participants to accelerate therapeutic development for pediatric-onset FSHD. The study aims to validate outcomes and refine clinical trial strategies. Previous cross-sectional studies suggest that younger age of onset is linked to greater clinical severity and that having 1-3 D4Z4 repeats is associated with extra-muscular complications in pediatric FSHD.

Prospective studies in early-onset FSHD have been limited by the small number of sites and low recruitment and follow-up rates. Early-onset pediatric FSHD is of high interest to drug companies because:

1. It results in a more significant disease burden than in adults.
2. Treating FSHD at earlier ages may have a more lasting and profound effect.
3. Genetic, molecular, and clinical factors may differ between pediatric and adult-onset FSHD.
4. Smaller body size and faster progression rates may make AAV-delivered gene therapies more feasible.

The FSHD CTRN's previous research showed that the FSHD composite functional measure (FSHD-COM), reachable workspace (RWS), and quantitative MRI measures (qMRI) are responsive to disease progression or treatment in adults with FSHD and correlate with performance. Investigators hypothesize that early changes in qMRI in pediatric subjects will predict 2-year changes in FSHD-COM Peds or RWS.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-17 years.
* Genetically confirmed FSHD (types 1 or 2).
* Symptomatic weakness (facial, shoulder, core, or limb weakness)
* Able to complete a 10-meter walk without the support of another person in less than 12 seconds (canes, walking sticks, and braces allowed; no walker). In order to include early onset participants up to 8 individuals will be entered with baseline 10MWR > 12 seconds or who are no longer ambulatory (≤10%)

Exclusion Criteria:

* Unwilling or unable to provide informed consent or assent. Any other medical condition which in the opinion of the investigator would interfere with study participation.
* Malignancy with ongoing treatment with chemotherapeutic agents or anabolic agents
* Use of immunosuppressants including prednisone or performance enhancing drugs including testosterone within 6 months
* Pregnancy
* Recent or ongoing infection
* Presence of contraindication to performance of MRI: pacemaker, metallic foreign body in eye, brain aneurysm clip (unless documented as MRI compatible)
* In the opinion of the investigator unable to follow directions for standardized testing

  * Note: Not being able to complete MRI will not result in a screen failure. If subject is not able to complete the procedure due to fear or anxiety, they will have the opportunity to try again at later visits. However, Subject must be willing to attempt to perform the MRI to meet inclusion/exclusion criteria

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is meant to target children most likely to be included in clinical trials: children who are clinically affected, old enough to perform functional measures, and still ambulatory. On outcomes proposed for MOVE Peds they would have room to show progression or improvement and be at a stage ideal to assess potential inclusion criteria: in particular whether symptom onset age or genetics separate early-onset from other childhood onset FSHD, or whether they exist on a spectrum of severities. At least half will qualify as early-onset (facial weakness before age 5 and shoulder weakness before age 10 or symptom onset before age 18 and 1-3 D4Z4 repeats). We will be also looking at a small cohort of early onset participants who's ambulation has been affected or is no longer able to ambulate. this will help us assess all child progression and understand the connection of early-onset and ambulation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Pediatric FSHD-COM | Baseline-2 years
  Investigators will collect the FSH-Composite outcome measure for children and adolescents. This measure assesses multiple body regions identified as important by patients, including leg function, shoulder and arm function, trunk function, hand function, and functional balance. The FSHD-COM Peds has been modified to include lighter weights for shoulder abduction and flexion, as well as elbow flexion, to accommodate the motor development and lower strength levels seen in children. Although the FSHD-COM Peds involves different measurements for each body region, these measurements are combined to produce a single composite score. The total score for the FSHD-COM Peds is out of 84, representing one comprehensive outcome measure
Reachable Work Space | Baseline-2 years
  Subjects are seated in front of a stereo-camera and perform a standardized upper extremity movement protocol under the supervision of a study clinical evaluator. Five-hundred-gram wrist weights will be added. The standardized simple set of movements consist of lifting the arm from the resting position to above the head while keeping the elbow extended, performing the same movement in vertical planes at around 0, 45, 90, 135 degrees. The second set of movements consists of horizontal sweeps at the level of the umbilicus and shoulder.

SECONDARY OUTCOMES:
Quantitative MRI (qMRI) Fat Fraction % | Baseline-2 years
  quantitative MRI measurements are considered gold standard for lean muscle volume measurement and disease biomarkers (fat volumes, fat faction, and STIR+ presence) that may be modulated by treatment. Muscle fat replacement and free-water hyperintensity indicate early disease changes before functional performance is affected. Muscles with an intermediate fat fraction (10-55%) predict disease progression over 1-2 years.
  Investigators will use a whole-body MRI and will find the fat fraction % in pediatric subjects and compare these measurements with other factors to create a composite score over a two-year period
Quantitative MRI (qMRI) Lean Muscle Volume (mL) | Baseline-2 years
  Quantitative MRI measurements are considered the gold standard for assessing lean muscle volume and disease biomarkers (fat volumes vs. lean muscle volumes and STIR+ presence) that may be modulated by treatment. Muscle fat replacement and free-water hyperintensity indicate early disease changes before functional performance is affected. Muscles with low lean muscle volume and an intermediate fat fraction (10-55%) predict disease progression over 1-2 years.
  Investigators will use whole-body MRI to measure lean muscle volume (mL) in pediatric subjects and compare these measurements with other factors to create a composite score over a two-year period.
Quantitative MRI (qMRI) Total Volume | Baseline-2 years
  Quantitative MRI measurements are considered the gold standard for assessing lean muscle volume and disease biomarkers (fat volumes, fat fraction and STIR+ presence) that may be modulated by treatment. The use of MRI has shown as a technique to predict disease progression.
  Investigators will use whole-body MRI to measure total volume (mL) in pediatric subjects and compare these measurements with other factors to create a composite score over a two-year period. This refers to the overall volume of a specific tissue or organ measured in milliliters (mL) using MRI.
Quantitative MRI (qMRI) STIR+ ( %) | Baseline-2 years
  Quantitative MRI measurements are considered the gold standard for assessing lean muscle volume and disease biomarkers, such as the percentage of lean muscle volume with Short Tau Inversion Recovery (STIR) enhancement. STIR MRI helps predict disease progression by highlighting areas of inflammation and edema within muscle tissue. This provides valuable insights into underlying disease processes, aiding in the prediction of progression and guiding treatment decisions.
  Investigators will use whole-body MRI to measure STIR positivity, indicating inflammation and edema, in pediatric subjects. These measurements will be compared with other factors to create a composite score over a two-year period.

OTHER OUTCOMES:
PROMIS Pediatric physical activity questionnaire (8 questions) | Baseline-2 years
  an instrument developed by the NIH PROMIS initiative. It generates scores for physical function and the impact of physical limitations on daily life. Participants will answer questions about how often they engage in physical activity, ranging from 0 days to 6-7 days per week. Higher scores indicate greater levels of physical activity.
Neuro Qol Fatigue Scale | Baseline-2 years
  assess the impact of fatigue on individuals with neurological conditions, measuring their severity, frequency, and effects on daily activities and quality of life using a 5- point rating system (1 being never and 5 being always).
The Facial Disability Index (FDI) physical score | Baseline-2 years
  is a 5-item questionnaire which assesses the physical impact of facial weakness. The responses (graded 1-5, 5 being no difficulty and 1 being unable to do) are summed to create a total score, which is then converted into a percentage scale. A score of 100% represents normal function, while lower scores indicate increasing levels of disability.
ACTIVLIM | Baseline-2 years
  measures how well people with neuromuscular disorders can perform daily activities. It includes 22 questions about tasks such as dressing, bathing, and walking, with difficulty rated as impossible, difficult, or easy.
Strength and Difficulties Questionnaire (SDQ) | Baseline-2 years
  is a tool used to screen for emotional and behavioral problems in children and adolescents aged 2 to 17. It consists of 25 questions divided into five categories: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Each item is rated on a 3-point scale (0= not true, 1 = somewhat true and 2 = certainly true)
Patient Global Impression of Severity (PGI-S) | Baseline-2 years
  Is a rating scale that patients can use to measure how severe they feel their symptoms are. Patients rate their condition on a scale from 1 (Normal) to 4 (Severe). This will serve as one of the study anchors.
Domain Delta | Baseline-2 years
  is an instrument developed to assess quality of life and how disease has changed since last visit. the purpose of the "domain-delta" questionnaire is to determine each patient's perceived change in their health-related quality-of-life in the last 6-months. This questionnaire will inquire about total health as well as health related to 14 subdomains self-identified as important by patients during development of the FSHD Health Index. Participants indicate their perceived change by answering if an area "is a lot worse", "is a little worse", "there has been no change", "it is a little better", or "it is a lot better" for each subdomain. This will serve as one of the other anchors in the study.
North Star Assessment for Dysferlinopathy (NSAD) | Baseline-2 years
  a tool used by clinicians to evaluate motor abilities in individuals with dysferlinopathy, a type of muscular dystrophy. It measures how well patients can perform various physical tasks, helping to track the progression of the disease. This assessment is useful for both walking and non-walking patients, providing important information to guide treatment and care plans. This will be used in comparison to how well the FSHD-COM Peds assessing subjects
Performance of Upper Limb (PUL) | Baseline-2 years
  an assessment tool used to evaluate upper limb function in individuals with muscular dystrophies, such as Duchenne muscular dystrophy. It measures the ability to perform various motor tasks, providing insights into the strength and mobility of the arms and hands. The PUL helps track disease progression and guides treatment decisions by capturing detailed information about upper limb capabilities. This will be helpful in assessing Cohort two as well as will be utilized to the FSHD-COM Peds and RWS.
100-Meter Walk/Run Test | Baseline-2 years
  is a fixed-distance assessment used to measure an individual's maximum ambulatory ability. Participants are asked to walk or run 100 meters as quickly as they can, depending on their capability. This test is commonly used in research to evaluate physical performance and mobility, particularly in individuals with conditions affecting their walking ability. It helps researchers track changes in mobility over time and assess the effectiveness of interventions aimed at improving walking speed and endurance
Neuro Qol Pain Scale | Baseline-2 years
  assess the impact of pain on individuals with neurological conditions, measuring their severity, frequency, and effects on daily activities and quality of life using a 5- point rating system (1 being never and 5 being always).
Patient Global Impression of Change (PGI-C) | Baseline-2 years
  Is a rating scale that patients can use to measure if any change in severity has occurred since being in the study. patient rate their change on a scale from 1 to 7 (1 being no change or worse and 7 being a great deal better or improvement that has made all the difference). This will serve as one of the study anchors.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center
Locations (7):
- United States (6):
  - Stanford University, Palo Alto, California
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah
- Murdoch Children's Research Institute, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No